CLINICAL TRIAL: NCT05311891
Title: Variants of SARS-CoV-2 in Central and West Africa: Frequency of Circulating Viruses and Implications for the Management and Control of the Pandemic
Brief Title: Variants of SARS-CoV-2 Causing COVID-19 in Africa
Acronym: South-Spike
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut de Recherche pour le Developpement (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS 0136s
Record Dates: First submitted 2022-03-23; First posted 2022-04-05 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Nasopharyngeal sample (virus)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective: 12000 participants positive for SARS-COV-2
  Interventions: Diagnostic Test: RT PCR
- Prospective: 600 participants positive for SARS-COV-2
  Interventions: Diagnostic Test: RT PCR

INTERVENTIONS:
Diagnostic Test: RT PCR — Characterize the different molecular variants of SARS-CoV-2, determine the escape potential of the new variants from neutralization by monoclonal antibodies and currently available vaccines and characterization of the mRNAs expressed in infected persons
  Other Names: Sequencing of the S gene; Sequencing of the entire SARS-COV-2 genome; Seroneutralization of antibodies; Respiratory transcriptomics

SUMMARY:
The main objective of this research is to identify and characterize the different molecular variants of SARS-CoV-2, emerging and / or circulating in several countries of Sub-Saharan Africa (Burkina Faso, Côte d'Ivoire, Gabon, Mali, Chad and Republic of Congo) and determine their role in the evolution of the pandemic.

DETAILED DESCRIPTION:
The main objective of this research is to identify and characterize the different molecular variants of SARS-CoV-2, emerging and / or circulating in several countries of Sub-Saharan Africa (Burkina Faso, Côte d'Ivoire, Gabon, Mali, Chad and Republic of Congo) and determine their role in the evolution of the pandemic.

The research will combine retrospective and prospective approaches to determine the evolutionary dynamics of the virus since the start of the pandemic. It is planned to sequence the entire Spike protein gene for 1550 viruses and make 300 entire genomes. This work will be supplemented by antibody seroneutralization and respiratory transcriptomics tests, in order to estimate the immuno-virological response of the COVID-19 disease associated with the identified SARS-CoV-2 variants.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (cf. country)
* Presenting for a SARS-COV-2 diagnosis, whether symptomatic or not
* Not objecting to participating in the research

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participant presenting for a SARS COV2 diagnosis, with or without symptoms
Sampling Method: Non-Probability Sample
Enrollment: 12600 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Number of SARS-CoV-2 sequences generated partially and in whole genome | Through study completion, an average of 1 year.
  This outcome represent our main gaol and will include sequences that were partially generated in the Spike proteine and full genomes as well. Our current target is 1550 sequences.

SECONDARY OUTCOMES:
Number of individuals tested positive for COVID-19 | Up to six months
  This outcome will be focused on the number of persons that will be tested positive for COVID-19 throughout the study, using SARS-CoV-2 rapid antigen tests. We planned to screen 12000 individuals overall in the six participating countries.
Number of new SARS-CoV-2 variants identify | Through study completion, an average of 1 year.
  This outcome represents the number of new viruses that are identified at the end of the study and have not been reported previously.

CONTACTS AND LOCATIONS:
Locations (6):
- Centre de Référence pour les pathogènes émergents et réémergent, Bobo-Dioulasso, Burkina Faso
- Centre Hospitalier Universitaire la Référence Nationale (CHU-RN), N'Djamena, Chad
- CIRBA, Abidjan, Côte d’Ivoire
- Unité Mixte de Recherche CIRMF-SSM, Libreville, Gabon
- SEREFO, Bamako, Mali
- Laboratoire National de Santé Publique Brazzaville, Brazzaville, Republic of the Congo